CLINICAL TRIAL: NCT01662843
Title: BRIPPED Scan for Evaluation of Emergency Department Patients With Shortness of Breath
Brief Title: BRIPPED Scan for Evaluation of Emergency Department (ED) Patients With Shortness of Breath
Acronym: BRIPPED
Status: Completed | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 11-07-FB-0204-HOSP
Record Dates: First submitted 2012-02-16; First posted 2012-08-10 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Dyspnea
Keywords: Dyspnea; Ultrasonography; Emergencies; Critical Care
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BRIPPED scan: Patients presenting with undifferentiated shortness of breath who receive the ultrasound scan in addition to standard of care
- Control: Patients who only receive the standard of care for undifferentiated shortness of breath

SUMMARY:
The B-RIPPED scan is a standardized ultrasound evaluation of pulmonary B-lines, Right ventricle size and strain, Inferior Vena Cava collapsibility, Pleural and Pericardial Effusion, Pneumothorax, Ejection Fraction, and lower extremity Deep Venous Thrombosis. Primary outcomes measured are the magnitude of change in differential diagnoses.

DETAILED DESCRIPTION:
This prospective randomized control trial will be performed on a convenience sample of 200 patients presenting with undifferentiated SOB to an academic emergency department (ED) (volume 56,000 patients/year). Subjects are excluded if they have a known history of asthma, are 20 or more weeks pregnant, or have had thoraco-abdominal trauma in the past 72 hours. The BRIPPED pilot investigation (IRB #10-02-FB-0026) enrolled 43 patients and physician subjects from 4/30/2010 to 1/20/2011. This study differs in methodology from the pilot study in the reduction of the total number of ultrasound images obtained to decrease the total time to perform the scan. Instead of a cohort study, this randomized control trial includes the addition of a control group for cost and time saved comparison. As in the pilot study, eligible patients will be evaluated by the treating ED physician who will rank potential diagnoses from most to least likely. A study investigator performs the B-RIPPED scan and provides the initial treating physician with the results. The treating physician will again be asked to complete a differential diagnosis ranking knowing the B-RIPPED results. Changes in the differential diagnosis ranking, physician orders, and interventions will be compiled. A randomized control cohort will be assigned for eligible patients. In the control group, the treating physician will complete the diagnosis rank list prior to the completion of the workup, and then once all lab values are back. Time to disposition, and comparison of labs and radiology tests ordered will be compared to the cohort receiving the BRIPPED scan. Patients will be assigned a number at time of enrollment, which randomly assigns them to the control or experimental (patients receiving the BRIPPED scan) group. Packets containing the appropriate data collection form (control or experimental) will be organized so even numbered patients will belong to one group, and odd numbered patients will be assigned to the other.

ELIGIBILITY:
Inclusion Criteria:

Subjects are included if they are between the ages of 18-89 and present to the Emergency Department with a chief complaint of shortness of breath or dyspnea.

Exclusion Criteria:

* known history of asthma,
* are 20 or more weeks pregnant, or
* have had thoraco-abdominal trauma in the past 72 hours.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of community subjects presenting to an Academic Hospital Emergency Department (volume approx 60,000 patients per year).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
magnitude of change of differential diagnosis of the treating physician | duration of ED course, which is expected to be an average of 3 hours

SECONDARY OUTCOMES:
time to complete the exam | 3 to 30 minutes during the ED course
time to disposition in control group compared to group receiving the BRIPPED scan | duration of ED course, which is expected to be an average of 3 hours, with a range of 45 minutes to 6 hours
labs, consults, medications and other orders added or discontinued after the treating physician is informed of the BRIPPED scan results | duration of the ED course, which is expected to be an average of 3 hours, with a range of 45 minutes to 6 hours
Recidivism rates among both cohorts, or evaluation of return to the ED within 30 days | 30 days after presentation to ED
  Electronic medical record review of patients who present with shortness of breath 30 days after initial presentation, evaluation and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Virginia M Stewart, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Sentara Norfolk General Emergency Department, Norfolk, Virginia, United States

REFERENCES:
- [Derived] Stewart VM, Bjornsson HM, Clinton M, Byars DV. BRIPPED scan for evaluation of ED patients with shortness of breath. Am J Emerg Med. 2016 Mar;34(3):386-91. doi: 10.1016/j.ajem.2015.11.006. Epub 2015 Nov 5. PMID 26704772